CLINICAL TRIAL: NCT03365908
Title: Pain Management of Anterior Cruciate Ligament Reconstruction: Evaluation of Adductor Canal Block Versus Oral Pain Regimen
Brief Title: Pain Management of ACL Reconstruction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1115203
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Operating surgeon and outcome assessor will be blind to whether patient had nerve block prior to OR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal Nerve Block (Experimental): Participant will receive an adductor canal nerve block via 15 mL 0.5% ropivacaine injection prior to OR for ACL reconstruction. Participant will receive pre-op oral medications.
  Interventions: Procedure: Adductor Canal Nerve Block; Drug: Ropivacaine injection
- No Nerve Block (No Intervention): Participant will receive pre-op oral medications but no nerve block prior to OR for ACL reconstruction.

INTERVENTIONS:
Procedure: Adductor Canal Nerve Block — An adductor canal nerve block with 15 mL of 0.5% ropivacaine will be performed pre-operatively by Anesthesiology.
  Arms: Adductor Canal Nerve Block
Drug: Ropivacaine injection — 15 mL of 0.5% ropivacaine will be administered for the adductor canal block
  Arms: Adductor Canal Nerve Block

SUMMARY:
This study will compare the outcome of pain interventions that are considered standard of care during the surgical treatment of ACL injuries. The comparison will be looking at pain control during and after ACL surgery as well as functional outcomes in patients that had a nerve block versus those who did not. The investigators hypothesize that pain control will be equal between both groups.

DETAILED DESCRIPTION:
Specific Aim #1: To determine if there is a difference in opioid pain medication use following anterior cruciate ligament (ACL) reconstruction between an oral pain regimen versus adductor canal block.

Specific Aim #2: To determine if there is a difference in knee recovery and function post-operatively following ACL reconstruction between an oral pain regimen versus adductor canal block.

Specific Aim #3: To determine if cost-effectiveness or patient flow logistics of ACL reconstruction are affected by whether has patient has adductor canal block versus receiving oral pain medication regimen.

Specific Aim #4: To determine if pre-operative Resiliency scores are associated with post-operative pain and outcomes following ACL reconstruction.

Hypothesis #1: There is no difference in post-operative pain management or functional outcomes following ACL reconstruction based on whether patient had adductor canal block versus an oral pain medication regiment implemented.

Hypothesis #2: Worse resiliency scores pre-operatively are associated with worse outcomes and pain scores post-operatively following ACL reconstruction.

Upon enrollment and at at the participant's pre-op appointment, the participant will complete a questionnaire entitled the Brief Resiliency Scale (BRS) to determine the participant's resiliency score and receive post-operative pain medication prescriptions. At time of surgery the participant will begin a pain diary to chronicle use of pain medication for 6 weeks and turn this document in at the 6-week follow-up appointment along with documentation of time to first able to walk (ambulate) without assistive device (i.e. crutch, walker, etc.). In the recovery room, the participant will verbally complete a Visual Analog Scale to determine the pain level at 15 minutes after surgery and before discharge. At the 3-month post-op visit, the participant will complete another questionnaire entitled the Knee Injury and Osteoarthritis Outcome Score (KOOS) to determine operative knee pain and function. At the 6-month post-op visit, the participant will complete a questionnaire entitled Marx Activity Rating Scale to determine operative knee function.

The treatment will be chosen by chance, like flipping a coin. Neither the participant nor the study doctor will choose what treatment the participant receives. The participant will have a one in two chance of being given each treatment. The participant will know which treatment was given but the operating surgeon will not know.

The participant will be randomized to 1 of 2 standard of care treatment groups at the time of surgery:

* Adductor canal nerve block (an anesthetic block of the femoral nerve halfway down the thigh that causes numbness in the knee and lower part of the leg)), or
* No nerve block for perioperative (during the operation) pain control.

Regardless of treatment group, all participants pre-operatively will receive the following pain medication: 400 mg celecoxib (Celebrex), 300 mg gabapentin (Neurontin), and 1 g of acetaminophen (Tylenol) 1-2 hours before surgery. This oral regimen is similar to standard of care pre-operative medication in total knee arthroplasties (knee replacements).

All participants will also receive the same post-operative prescriptions at their pre-operative clinic visit which will be: 90 tablets of 1 g acetaminophen to be taken three times a day for 30 days and 90 tablets of 5 mg oxycodone with 1-2 tablets to be taken every 4 to 6 hours as needed for pain. Additionally, the participant will receive two medications (Zofran, Phenergan) for nausea/vomiting which are to be taken as needed. Participants will record their medication use.

ACL reconstruction and any other procedures to address any other damage in the participants's knee as determined by the surgeon will be performed as per standard clinical practice at an outpatient surgical facility. The participant will undergo standard post-operative rehabilitation. During the standard of care post-operative visits in the Sports Medicine Clinic, the participant will be asked to fill out questionnaires specific for our data collection.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45 years old.
* Clinical and/or advanced imaging confirmation of ACL tear of which reconstructive surgery is recommended and accepted.

Exclusion Criteria:

* No prior surgery of the affected and contralateral knee
* Adults unable to consent
* Children (age < 18 years old)
* Prisoners
* Pregnant women
* Inflammatory arthritis
* Non-English-speaking patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Immediate Post-op Pain Score | 15 min post-op
  Measured via Visual Analog Scale (VAS) in recovery, scale from 0 (least) to 10 (maximum), no units, with 0 being no pain and 10 being extreme pain
Opioid Use | 6 weeks post-op
  Aggregated amount of narcotic medication used, measured in milligrams

SECONDARY OUTCOMES:
Short-term Knee Function Post-op | 6 weeks post-op
  Functional recovery of knee following surgery as measured by Knee Injury and Osteoarthritis Outcome Score (no units), range from 0 - 100 with 0 representing extreme problems with the knee and 100 representing no problems
Intermediate-term Knee Function | 12 weeks post-op
  Functional recovery of knee following surgery as measured by Marx activity score (no unit), 0 - 16, with 0 representing significant limitation in activity due to knee and 16 representing no limitations
Long-term Knee Function | 24 weeks post-op
  Functional recovery of knee following surgery as measured by Tegner activity score (no units), range from 0 - 10, with 0 representing inability to work or perform daily activities due to knee and 10 representing ability to compete in high-level activities
Post-anaesthesia care unit (PACU) Time | Immediately after surgery
  Amount of time, measured in minutes, participants required in PACU before discharge due to pain control

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Lee, MD, Principal Investigator — UC-Davis Health
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronowitz ER, Kleinbart FA. Outpatient ACL reconstruction using intraoperative local analgesia and oral postoperative pain medication. Orthopedics. 1998 Jul;21(7):781-4. doi: 10.3928/0147-7447-19980701-07. PMID 9672915
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- See also: Learn more or sign up for the study here! — https://studypages.com/s/pain-management-after-acl-reconstruction-surgery-952138/